CLINICAL TRIAL: NCT05315089
Title: Effects and Perception of Intensive Virtual Reality Training on Upper Limb Functions After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/01245 Iqra Butt
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Stroke
Keywords: intensive virtual reality; upper limb functions
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): Virtual reality games +conventional exercises
  Interventions: Other: Virtual reality games +conventional exercises
- control Group (Active Comparator): Conventional exercises
  Interventions: Other: Conventional exercises

INTERVENTIONS:
Other: Virtual reality games +conventional exercises — Virtual reality games +conventional exercises
  Arms: Interventional Group
Other: Conventional exercises — Conventional exercises
  Arms: control Group

SUMMARY:
Previous literature review shows limited work on upper limb recovery from Virtual Reality device and most of them are pilot studies meta-analysis some Randomized control Trial studies are done but this study will cover mixed method including both qualitative and quantitative method.

DETAILED DESCRIPTION:
Stroke is the leading cause of disability worldwide Approximately 80% of stroke survivors regain ability to walk, 30 - 66% of survivors are not able to use their affected upper limb mobility. With improving survival rates and longer life expectancy in general, the burden of caring for stroke survivors is likely to increase. As a lack of upper limb recovery results in significant dependence and a reduced quality of life. Persistent upper limb (UL) dysfunction after a stroke is one of the most challenging issues in rehabilitation. Effective upper limb treatment interventions have therefore been identified as a priority for stroke research. One of the rehabilitation strategies include performing self-administered exercises using VR games technology. Effective treatment interventions post-stroke is characterized by high intensity and repetitive practice of a meaningful task. However, changes in infrastructure, an emphasis on mobility during early rehabilitation ,to reduce hospital length of stay and a lack of therapy on discharge home have resulted in challenges delivering the amount of rehabilitation necessary to optimize recovery. A promising technique, which has the capability of creating an interactive environment in which practice intensity and feedback can be manipulated to retrain movement in the upper limb in people with stroke, is virtual reality (VR) technology .VR provides a sense of illusion: of being immersed in a world where objects can he visualized and interact with. The system is usually a controlled one, where the objects and interaction styles (point, touch, grasp) are defined prior to the controlling program being executed. There are a number of ways in which the virtual environment (VE) can he presented to the user. Most common are desktop (fish tank) VR systems where the VE is displayed on a standard desktop monitor. The user can interact with the environment via standard hardware (keyboard, mouse) or via specialized VR devices such as data gloves, hut is conscious of 'looking at' the environment rather than 'immersed in' the environment.

ELIGIBILITY:
Inclusion Criteria:

1- Subacute and chronic stroke patient > 3 months post stroke till 1 year. 2. Both gender 3. Age: 40-70 years 4. Modified Ashworth scale1-3 5. MMSE>25 6. Able to follow verbal instructions related to the use of VR devices

Exclusion Criteria:

1. Neurological disorders other than stroke.
2. Aphasia that would limit the ability to follow verbal instructions.
3. Participation in other upper extremity therapies during the study

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Fugl- Meyer assessment upper extremity | Change from Baseline , motor functions to 3 Week, to 6 week
  The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia
Chedoke Arm and Hand Inventory | Change from Baseline , motor functions of hand to 3 Week, to 6 week
  The Chedoke Arm and Hand Activity Inventory (CAHAI) is a functional assessment of the recovering arm and hand after stroke

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, MSNMPT, Principal Investigator — Riphah college of Rehabilitation and Allied Health sciences Islamabad
Locations (1):
- Misbah Ghous, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hughes AM, Burridge JH, Demain SH, Ellis-Hill C, Meagher C, Tedesco-Triccas L, Turk R, Swain I. Translation of evidence-based Assistive Technologies into stroke rehabilitation: users' perceptions of the barriers and opportunities. BMC Health Serv Res. 2014 Mar 12;14:124. doi: 10.1186/1472-6963-14-124. PMID 24620739
- [Background] Ward N, Kelly K, Brander F. The future of stroke rehabilitation: upper limb recovery. ACNR. 2015;15(4):6-8.
- [Background] Elnady A, Mortenson WB, Menon C. Perceptions of Existing Wearable Robotic Devices for Upper Extremity and Suggestions for Their Development: Findings From Therapists and People With Stroke. JMIR Rehabil Assist Technol. 2018 May 15;5(1):e12. doi: 10.2196/rehab.9535. PMID 29764799
- [Background] Lohse KR, Hilderman CG, Cheung KL, Tatla S, Van der Loos HF. Virtual reality therapy for adults post-stroke: a systematic review and meta-analysis exploring virtual environments and commercial games in therapy. PLoS One. 2014 Mar 28;9(3):e93318. doi: 10.1371/journal.pone.0093318. eCollection 2014. PMID 24681826